CLINICAL TRIAL: NCT04981951
Title: Dexmedetomidine as an Adjuvant to Local Anesthesia in Supraclavicular Plexus Block, A Randomized Control Trial.
Brief Title: Th Effects of a Drug Dexmedotemidine in Regional Anesthesia in Participants Undergoing Upper Limb Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zaher Nazzal (Other)
Responsible Party: Sponsor-Investigator, Zaher Nazzal, Head of Research Unit, An-Najah National University
Organization: An-Najah National University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: F.Med.25th August/2020/10
Record Dates: First submitted 2021-05-30; First posted 2021-07-29 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Supraclavicular Brachial Plexus Block
Keywords: Dexmedetomidine; Randomized Controlled Trial.; Supraclavicular Plexus Block; bupivacaine; Palestine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine and Bupivacaine (Experimental): Patients will be given Dexemtomidine ( the intervention) added to the Bupivacaine
  Interventions: Drug: Dexmedetomidine
- Bupivacaine alone (No Intervention): patients will be given Bupivacaine alone

INTERVENTIONS:
Drug: Dexmedetomidine — Highly selective α2-adrenergic receptor agonist. With sedative, analgesic, peri-operative sympatholytic and hemodynamic stabilizing properties.
  Other Names: non
  Arms: Dexmedetomidine and Bupivacaine

SUMMARY:
In this study, we will assess the effect of combined Dexmedetomidine and Bupivacaine analgesia on the onset and duration of anesthesia in supraclavicular plexus block compared to Bupivacaine alone.

DETAILED DESCRIPTION:
Participants who fulfill the inclusion criteria will be enrolled in this study to achieve sample size of 140 participants, 70 participants in each group.

Participants were blindly randomized into two groups: group A (Bupivacaine alone) and group B (Bupivacaine with Dexmedetomidine).

On the morning of the surgery day, and before performing the procedure on the targeted hand, a venous cannula 18gauze was secured on the opposite hand. Routine monitors like pulse oximetry, non-invasive blood pressure, and electrocardiogram were attached during the procedure.

Study medications were prepared for each group, which is Bupivacaine (30ml) only for group A and Bupivacaine (30 ml) with Dexmedetomidine (1 mcg /kg) for group B. Then, SCPB was done under ultrasound guidance which increases the safety due to improved monitoring of anatomy and needle placement. A needle was placed within the brachial plexus sheath posterior to the subclavian artery, and the local anesthetic injected to surround the trunks and divisions of the brachial plexus at this level.

Patients were evaluated for the onset of the sensory and motor block every 3 minutes after completion of injection till their onset, and, at 15, 30, 45, 60, 90, and 120 min; and then hourly (even after surgery), until they had resolved.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-75 years.
* Classified as grades 1 or 2 by the American Society of Anesthesiology Classification of .physical status.
* Willing and able to sign a consent form.

Exclusion Criteria:

* Patients under the following conditions will be excluded: Known hypersensitivity to Bupivacaine, Dexmedetomidine, and local anesthetics.
* Uncontrolled diabetes mellitus.
* Peripheral neuropathy.
* SevereCoagulopathy.
* Infection at the site of block.
* Pregnancy.
* Cardiac arrhythmias.
* Prescription of beta blockers.
* Psychological disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
The onset of anaesthesia in supraclavicular plexus block | "up to 9 hours"
  Sensory block assessed by pinprick test with a blunt 25-G hypodermic needle. Grade 0: sharp pin sensation felt, grade 1: analgesia, dull sensation felt, grade 2: anesthesia, no sensation felt the onset of sensory block is the interval between the end of total local anesthetic administration and sensory block grade 1
The duration of anesthesia in supraclavicular plexus block | "up to 9 hours"
  The motor blockade assessed using the Modified Bromage scale (MBS). Grade 0: able to raise the extended arm to 90 degrees for 2 seconds; grade 1: able to bend the elbow and move the fingers but not the extended arm; grade 2: unable to flex the elbow but able to move the fingers; grade 3: unable to move the arm, elbow, and fingers. The onset of the motor blockade is the interval from injection of the local anesthetic to motor analysis equivalent to Bromage score 2

SECONDARY OUTCOMES:
Intraoperative heart rate | "1 hour"
  Heart rate per min is assessed intraoperatively
Intraoperative blood pressure as mm Hg | "1 hour"
  Blood pressure assessed by a non-invasive monitor
Intraoperative somnolence | "1 hour"
  Somnolence assessed using Ramsay Sedation Scale. It grades somnolence on a scale of 1-6: 1 = anxious, agitated, restless; 2 = cooperative, oriented, tranquil; 3 = responds to commands only; 4 = brisk response to light glabellar tap or loud noise; 5 = sluggish response to light glabellar tap or loud noise; 6 = no response
Post-operative heart rate | "up to 6 hours"
  Heart rate per min is assessed postoperatively
Post-operative blood pressure | "up to 6 hours"
  Blood pressure assessed by a non-invasive monitor
Post-operative somnolence | "up to 6 hours"
  Somnolence assessed using Ramsay Sedation Scale. It grades somnolence on a scale of 1-6: 1 = anxious, agitated, restless; 2 = cooperative, oriented, tranquil; 3 = responds to commands only; 4 = brisk response to light glabellar tap or loud noise; 5 = sluggish response to light glabellar tap or loud noise; 6 = no response
Number of Participants With Postoperative nausea and vomiting. | "up to 6 hours"
  Vomiting assessed by mentoring the patients actively. Nausea assessed by asking the patients directly.

CONTACTS AND LOCATIONS:
Overall Officials: Zaher Nazzal, MD, Principal Investigator — An-Najah National University; Wael Sadaqa, MD, Study Director — An-Najah National University
Locations (1):
- Zaher Nazzal, Nablus, Wes-Bank, Palestinian Territories